CLINICAL TRIAL: NCT04972747
Title: SBÜ Koceli Derince Eğitim ve Araştırma Hastanesi
Brief Title: The Effect of Skin Care Applied With Two Different Oils on Skin Integrity and Growth Parameters in Premature Babies
Acronym: DEAH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Derince Training and Research Hospital (Other)
Collaborators: Okan University (Other)
Responsible Party: Principal Investigator, Yaprak Tokdemir, Principal Investigator, Derince Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2020/124-2
Record Dates: First submitted 2021-05-20; First posted 2021-07-22 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Premature Birth; Skin Care
Keywords: skin care; preterm; coconut oil; sunflowers oil; growth parameter
MeSH Terms: conditions — Premature Birth | interventions — Skin Care; Sunflower Oil; Coconut Oil

STUDY DESIGN:
Intervention Model Description: randomized controlled clinical trial
Who Masked: Investigator
Masking Description: Babies meeting the criteria will be divided into two groups by randomization method. Randomization will be done by drawing lots using two red and blue cards. 31 red and 31 blue cards will be placed in an invisible purse. For the baby who meets the criteria, a card will be drawn by another nurse working in the clinic. Massage with sunflower oil will be applied for the baby with a red card, and skin care with coconut oil will be applied for the baby with a blue card.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Suggest skin care with sunflower oil for preterm babies (Experimental): * Before each application, preterm babies will be given skin care in the service routine and sunflower oil will be applied twice a day for 14 days.
  * Absorption of sunflower oil for preterm babies will be provided by using a baby massage application.
  * Before the massage, 3-4 ml of sunflower oil will be applied to the whole body surface except the genital area and scalp..
  * 12 hours after each application, the skin of the newborn will be evaluated using the "Neonatal Skin Condition Assessment Scale" (Appendix-2), and the measurement will be made with a DMM brand skin moisture meter and recorded in the follow-up form.
  Interventions: Other: skin care with sunflower oil
- Suggest skin care with cocunut oil for preterm babies (Experimental): * Before each application, preterm babies will be given skin care in the service routine and coconut oil will be applied twice a day for 14 days.
  * Absorption of coconut oil for preterm babies will be provided by using a baby massage application.
  * Before the massage, 3-4 ml of coconut oil will be applied to the whole body surface except the genital area and scalp.
  * 12 hours after each application, the skin of the newborn will be evaluated using the "Neonatal Skin Condition Assessment Scale" (Appendix-2), and the measurement will be made with a DMM brand skin moisture meter and recorded in the follow-up form.
  Interventions: Other: skin care with sunflower oil

INTERVENTIONS:
Other: skin care with sunflower oil — The application will be carried out twice a day during the maintenance hours of the service. In skin care applications, body baths are applied not more than three times a week, as it may cause hypothermia in preterm babies in the ward routine. In daily skin care, body cleaning with cotton, changing the fixation points such as orogastric probe, and changing the monitor probe locations are among the routine practices. In order to hydrate and moisturize the skin in preterm and term babies, baby oil in the service is used. Skin care applied in the service routine will be applied to the preterm babies included in the study, and only sunflower oil and coconut oil will be used as moisturizers.
  Other Names: skin care with coconut oil

SUMMARY:
As a result of technological advances in the field of newborns, the survival rates of very young babies have increased. With this situation, there was a need to develop new evidence-based application areas in premature babies. Nurses provide evidence-based care in many areas to term and preterm babies in the neonatal intensive care unit. One of these areas is the skin, which is known as 13% of the newborn's body weight and constitutes the largest part of the organism. Before skin care is given, knowing the skin characteristics of the newborn and performing skin care in accordance with these features will provide more benefits for the baby. The skin of newborns is different from adults in terms of both function and function. In addition, skin characteristics of term and preterm babies also differ according to the week of delivery.

Skin basically enables the newborn to explore the world by thermoregulation, as a barrier against microorganisms and chemical harmful substances, maintaining fluid-electrolyte balance, vitamin D production, fat storage and sensory-touch. The immature skin of the newborn cannot fully fulfill these functions. In another study conducted between sunflower oil and the control group, it was stated that rash and peeling were less common in the sunflower oil experiment group compared to the control group.

As a result, evidence-based knowledge of nurses about neonatal skin care should be increased in neonatal intensive care units, and appropriate nursing care should be given especially to premature newborns who are at risk due to hospitalization. Even if there is no routine procedure in our service, baby oil is massaged during care hours, but there is no study on this. The aim of this study is to contribute to the neonatal skin care literature and to provide appropriate evidence-based care in the service routine.

DETAILED DESCRIPTION:
The research will be carried out with preterm babies hospitalized in the 3rd Level Neonatal Intensive Care Unit of SBÜ Kocaeli Derince Training and Research Hospital, Alikahya Campus and meeting the criteria of the study. Preterm babies with a birth weight of 1000 g and above, who do not receive ventilator support, and who do not have skin damage more than 5% of the body surface between 32-36 weeks of gestation will be included in the study. Two groups will be created by randomization method.

These groups are; Sunflower oil group: Babies to whom skin care will be applied with sunflower oil.

Coconut oil group: Babies who will be treated with coconut oil

After the premature babies who meet the study criteria are divided into groups and their consent is obtained, they will be followed up by the person conducting the study, and all applications will be carried out by the same person. Information about the newborn will be filled in by the person who will perform the application by using the "Form for Identifying the Introductory and Clinical Characteristics of the Newborn".

The application will be carried out twice a day during the maintenance hours of the service. In skin care applications, body baths are applied not more than three times a week, as it may cause hypothermia in preterm babies in the ward routine. In daily skin care, body cleaning with cotton, changing the fixation points such as orogastric probe, and changing the monitor probe locations are among the routine practices. In order to hydrate and moisturize the skin in preterm and term babies, baby oil in the service is used. Skin care applied in the service routine will be applied to the preterm babies included in the study, and only sunflower oil and coconut oil will be used as moisturizers.

APPLICATION Group 1: Preterm babies treated with sunflower oil

* 31 preterm babies determined by randomization method will be included in the group to be applied skin care with sunflower oil.
* Before the application, the researcher will meet with the family and fill in the "Informed Consent Form".
* Social hand washing will be applied before the application.
* Before the application, the skin of the newborn will be evaluated by using the "Neonatal Skin Condition Assessment Scale".
* In order to measure the moisture of the skin before the application, the moisture level of the skin will be recorded by measuring from three different points, namely the abdomen, legs and arms, with a DMM branded skin moisture meter.
* The baby will be placed under a radiant warmer by the practitioner to keep his body temperature.
* For the follow-up of growth parameters, the weight of the newborn will be weighed at the same time while the baby is naked, using the digital baby scale in the service. In addition, the baby's head circumference, height and belly circumference will be measured with a tape measure and recorded.
* Before each application, preterm babies will be given skin care in the service routine and sunflower oil will be applied twice a day for 14 days.
* Absorption of sunflower oil for preterm babies will be provided by using a baby massage application.
* Before the massage, 3-4 ml of sunflower oil will be applied to the whole body surface except the genital area and scalp.
* Massage to the baby will be started first on the legs and feet, then continued with massage of the abdomen and chest area, arms and hands, face and back, respectively, and will be applied for 15 minutes at least 30 minutes after feeding.
* 12 hours after each application, the skin of the newborn will be evaluated using the "Neonatal Skin Condition Assessment Scale", and the measurement will be made with a DMM brand skin moisture meter and recorded in the follow-up form.
* Weight monitoring will be recorded daily to monitor growth parameters and daily weight gain / decrease will be monitored. Head circumference and height lengths will be measured and recorded before the application and on the 7th and 14th day of the application.

Group 2: Preterm babies treated with coconut oil

* 31 preterm coconut oils determined by randomization method will be included in the group to be applied skin care.
* Before the application, the researcher will meet with the family and fill in the "Informed Consent Form".
* Social hand washing will be applied before the application.
* Before the application, the skin of the newborn will be evaluated by using the "Neonatal Skin Condition Assessment Scale".
* In order to measure the moisture of the skin before the application, the moisture level of the skin will be recorded by measuring from three different points, namely the abdomen, legs and arms, with a DMM branded skin moisture meter.
* The baby will be placed under a radiant warmer by the practitioner to keep his body temperature.
* For the follow-up of growth parameters, the weight of the newborn will be weighed at the same time while the baby is naked, using the digital baby scale in the service. In addition, the baby's head circumference, height and belly circumference will be measured with a tape measure and recorded.
* Before each application, preterm babies will be given skin care in the service routine and coconut oil will be applied twice a day for 14 days.
* Absorption of coconut oil for preterm babies will be provided by using a baby massage application.
* Before the massage, 3-4 ml of coconut oil will be applied to the whole body surface except the genital area and scalp.
* Massage to the baby will be started first on the legs and feet, then continued with massage of the abdomen and chest area, arms and hands, face and back, respectively, and will be applied for 15 minutes at least 30 minutes after feeding.
* 12 hours after each application, the skin of the newborn will be evaluated using the "Neonatal Skin Condition Assessment Scale", and the measurement will be made with a DMM brand skin moisture meter and recorded in the follow-up form.
* Weight monitoring will be recorded daily to monitor growth parameters and daily weight gain / decrease will be monitored. Head circumference and height lengths will be measured and recorded before the application and on the 7th and 14th day of the application.

Sunflower oil

Sunflower oil is a light yellow colored and light-tasting vegetable oil obtained from the seeds of the sunflower plant. It contains 90% unsaturated fatty acids (combined oleic and linoleic) and about 10% saturated fatty acids (palmitic and stearic). In the literature, the importance of using mineral oils in maintaining the integrity of the skin of newborns has been stated and there are many studies using sunflower oil on this subject.

Coconut Oil

Coconut oil is a highly saturated fat traditionally made from the oil's raw coconut or dried coconut kernels. Coconut oil is rich in medium-chain fatty acids, a saturated form of fat. It contains Lauric acid 49%, Mystic acid 18%, Caprylic acid 8%, Palmitic acid 8% and Capric acid 7%.

Recruitment Criteria;

* Parents' consent to participate in the research
* Preterm babies at 32-36 gestational week
* preterm babies with a weight of 1000 gr and above
* Non-surgical infants are included

Exclusion Criteria;

* Preterm babies monitored on mechanical ventilation
* Skin damage over 5% of the body surface
* Preterm babies receiving phototherapy

ELIGIBILITY:
Inclusion Criteria:

* Parents' agreement to participate in the research
* Preterm babies at 32-36 gestational week
* 1000 gr and above preterm babies
* Non-surgical infants are included.

Exclusion Criteria:

* Skin damage may occur over 5% of the body surface
* Preterm babies monitored on mechanical ventilation
* Preterm babies receiving phototherapy

Ages: 2 Days to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
The effect of skin care applied with two different oils on skin integrity and growth parameters in premature babies | one year
  Neonatal Skin Condition Score-NSCS. The scale consists of three parameters. These; dryness, redness and deterioration of skin integrity/peeling. Each parameter is scored from one to three. The lowest score that can be obtained from the scale is 3, the highest score is 9, and a total score of 16 indicates that the skin condition of the newborn is poor.

CONTACTS AND LOCATIONS:
Overall Officials: Gülzade Uysal, assoc. prof, Principal Investigator — Okan University
Locations (1):
- Derince eğitim ve Araştırma Hastanesi, Kocaeli, İ̇zmi̇t, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No